CLINICAL TRIAL: NCT04187729
Title: Intermountain Healthcare's - PRECISion MEdicine Biobank
Brief Title: Precision Genomics Medicine Biobank
Acronym: PRECISE
Status: Recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Tyler Barker, PhD, Senior Scientist, Intermountain Health Care, Inc.
Other Study IDs: 1050678
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Any Disease Condition and Reportedly-healthy Subjects

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased: Subjects with a known disease.
- Non-diseased: Subjects without a known disease and reportedly healthy.

SUMMARY:
The immediate goal of this study is to collect biological samples (i.e., tissue and/or fluid), clinical information, and laboratory data from disease and non-disease subjects seen at Intermountain Healthcare affiliated facilities. The long-term goal is to annotate tissue and/or fluid biomarker data to clinical information and laboratory data for the purpose of improving health care delivery and prognostic potential.

DETAILED DESCRIPTION:
This study consists of an observational, non-randomized, open, long-term study in diseased and non-diseased subjects. There are no investigational treatments, drugs, or procedures associated with subject participation. This study will consist of two groups:

1. Group #1: Diseased subjects (including COVID-19 known positive subjects)
2. Group #2: Non-diseased subjects

   The biological samples collected may be tested numerous times for genes/biomarkers, and not yet-discovered genes/biomarkers, and other genetic and biological materials associated with healthcare-related conditions. In some cases, cells or tissues may be maintained in culture in order to study functions of living cells in both a healthy and diseased state.

   Disease subjects who qualify for this project (see inclusion and exclusion criteria) will continue with their usual or specialized care for their underlying health-care related condition(s).

   Disease subjects (Group #1)

   Other than the visit(s) for obtaining informed consent, the collection of biological samples, and the hand dynamometer test, subjects will have no other responsibilities to this project with regard to additional or follow-up visits, however sample collection may continue at routine standard of care visits. The collection and storage of tissue and/or fluid will be as the following:
   * The storage of tissue or fluid that is collected during a routine, standard of care procedure(s) or treatment(s) that is leftover following clinical testing or is otherwise discarded,
   * The storage of blood collected as a stand-alone blood draw procedure or during a routine, standard of care blood draw procedure,
   * The storage of tissue or fluid that is collected separate from standard of care procedures, such as a blood draw and/or buccal swab, and/or
   * The storage of additional tissue or fluid that is collected during a routine, standard of care image guided biopsy (for example, collection of additional tumor samples during a computed tomography guided biopsy) under the direction and discretion of the interventional physician. Additional biopsies will be limited up to 4 cores with the size of each core biopsy being equivalent to a grain of rice.

   Biological samples will be collected as appropriate, based on the subject's underlying healthcare related condition, either during a routine or specialized care procedure, when other ordered lab work is done, or as a stand-alone sample collection. Participating subjects may be asked to provide consent to one or more collections of biological samples. Biological sample collection from the general population subjects may be a separate blood draw and/or buccal swab.

   Examples of the biological samples that may be collected are as follows (but not limited to):
   * Blood/Plasma (up to 40 ml of blood)
   * Ascites
   * Bone Marrow
   * Buccal smear (cheek)
   * Cartilage
   * Cerebrospinal fluid
   * Mucus
   * Saliva
   * Sputum
   * Stool
   * Sweat
   * Synovial fluid
   * Tears
   * Tissue samples (e.g. muscle, skin, nails, tumor, etc.)
   * Urine
   * Seminal fluid
   * Genetic material extracted from any biological sample
   * Other biological samples as identified by the Principal Investigator or Co-Investigators and agreed by the subject

   Buccal swab will be an alternative source of DNA when blood or other biological samples cannot be obtained. In some instances, the remaining portion of specimens obtained for diagnostic purposes will be used. The use of these residual clinical specimens may sometimes (but not always) make the collection of a blood specimen by venipuncture unnecessary.

   Prior to each blood draw (i.e., at stand alone or part of standard of care if the investigators are performing the blood draw), or other biological sample collection, subjects will perform 3 maximal effort handgrip strength tests. In a seated position with the elbow bent to 90 degrees of flexion, each contraction will be 3 seconds in duration. Contractions will be separated by 60 seconds of rests. All contractions will be performed by the patients-reported dominant hand. The investigators will record the peak force from each contraction.

   Patients that have been previously tested for COVID-19 will be uniquely handled. Specifically, Intermountain Healthcare patients previously tested and with a known positive or negative COVID-19 result available in the Intermountain Healthcare electronic medical records will be recruited for study participation. Subjects will undergo a remote phone script electronic consent procedures for the purpose of collecting saliva.

   Saliva samples will be collected once in each subject at the Intermountain Healthcare locations identified below. It is possible, however, that a second sample may be needed. Reason for the collection of a second saliva sample may include, but is not limited to: confirmational testing of the first sample, the first sample was inadvertently compromised or destroyed, or for other unforeseeable reasons, such as virus exposure after the initial sample was collected. Subjects that consented to this study may provide an additional sample(s) for up to 1-year after enrollment if they feel like they have been in contact or exposed to COVID-19. Approximately 2.0 mL of saliva will be collected with each saliva kit.

   Saliva collection kits (see below for description) for Intermountain Healthcare providers will be available for pick-up at the following sites:
   * COVID-19 screening location on the Dixie Regional Medical Center campus,
   * Primary Outpatient Laboratory at Dixie Regional Medical Center,
   * Dixie Regional Cancer Center Laboratory, and
   * Eccles Outpatient Laboratory Intermountain Medical Center (Murray, UT)

   Saliva samples will be dropped-off at the location where the kits are available. Kits are not required to be dropped-off at the same location as pick-up. When necessary, saliva kits will be mailed to subjects with the appropriate material for an expedited return to Precision Genomics at the Intermountain Healthcare - Cancer Center (St. George, UT). Saliva samples may be obtained during the caregivers' routine shift (preferably at the end of their shift).

   Saliva will be collected using a self-collection kit (Zymo Research, Irvin, CA USA, catalog #: R1210) that provides the materials and instructions for collecting and stabilizing the specimens. We anticipate sample collection to take 2 to 5 minutes. After collection, saliva samples will be sent or delivered to the Intermountain Healthcare Cancer Center (St. George, UT). Samples will be immediately de-identified.

   Saliva samples will be tested for the presence of COVID-19 using a previously published rtPCR-based protocol to specifically detect COVID-19 RNA at Precision Genomics (Intermountain Healthcare, Cancer Center, St. George, UT USA). Saliva samples may also undergo various genotyping, whole genome sequencing, transcriptomic interrogation, and proteomic analyses, and may be tested numerous times for genomic and/or genetic biomarkers, and not-yet-discovered genes/biomarkers, and other genetic and biological materials associated with healthcare-related conditions in other follow-up studies.

   Although we anticipate utilizing the procedures described above, the challenges associated with this novel virus may require the necessity of implementing a variety of different assays and procedures to develop a robust and valid testing procedure. Therefore, it is plausible that DNA will be analyzed by downstream molecular technologies, such as next-generation sequencing, digital drop polymerase chain reaction (ddPCR), and other proteomic and molecular analyses. With that said, all data analyses and analytical procedures will be performed at Intermountain Healthcare's - Precision Genomics.

   Negative results will not be returned to subjects. In the case of a positive research-based test result, a clinical research coordinator will contact and direct the participant to obtain another COVID-19 test at participating Intermountain Healthcare COVID-19 testing sites. We expect results from the research-based screening test to be returned within 24-hours.

   Although not likely, there is a possibility that an Intermountain Healthcare patient with a previously known negative test could test positive with the COVID-19 testing performed with participation in this study. In this situation, the subject will be informed of the new positive test result and immediately advised to seek conformational testing at a nearby COVID-19 screening location.

   DNA extraction from the biological samples will be performed and stored at the Translational Science Center in St. George, UT USA. For novel disease-causing gene searches that may be done, biological samples will be sent to collaborating laboratories and/or organizations, depending on the needed specialty and the likelihood of finding a novel gene. If researchers or the consulting laboratory require additional information in order to perform phenotype/genotype correlation studies, results from tests such as standard physical examinations may be requested. These tests will be requested and/or conducted through the subject's primary care physician.

   Non-disease subjects (Group #2)

   Other than the visit for obtaining informed consent, the collection of biological samples, and the hand dynamometer test, subjects will have no other responsibilities to this project with regard to additional or follow-up visits, however sample collection may continue at routine standard of care visits. The collection and storage of tissue and/or fluid will be as the following:
   * The storage of tissue or fluid that is collected during an elective-surgical procedure (such as anterior cruciate ligament surgery) that is otherwise discarded, and/or
   * The storage of tissue or fluid that is collected separate from standard of care procedures, such as an elective and consented blood draw and/or buccal swab procedure for the storage and use of the subject's blood for various analytical procedures.

   Study duration

   There is no planned end-date for this project; therefore, the study duration is indefinite for the recruitment of subjects, collection of biological samples, and/or for completion of the project. All biological samples collected and patient information obtained will be archived in long-term storage at an Intermountain Healthcare facility.

   Subjects may be screened at all participating facilities within Intermountain Healthcare.

   Following screening and recruitment into the project, and after samples are obtained, participating subjects will not have any other follow up or non-standard of care visits required by this project, however sample collection may continue at routine standard of care visits. For this project, subjects give consent for unrestricted use of his/her sample(s), i.e. the sample(s) will be used indefinitely, until it is gone or until the patient withdraws consent.

   Study enrollment

   Enrollment is open-ended in this study, and therefore, there is no planned targeted enrollment accrual.

ELIGIBILITY:
Group #1 inclusion criteria

* Male and female adults (≥ 18 years of age)
* Diagnosed with any healthcare-related condition(s)
* Subject presenting to an Intermountain Healthcare facility

Group #2 inclusion criteria

* Male and female adults (≥ 18 years of age)
* Reportedly healthy (i.e., non-diseased)
* Subject presenting to an Intermountain Healthcare facility

Groups #1 and 2 exclusion criteria

* Inability or refusal of the patient and/or the patient's legally-acceptable representative to provide informed consent for any reason
* Other conditions that the Principal Investigators or Co-Investigators believe may increase the risk to the subject and/or compromise the scientific integrity of the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any subject (i.e., diseased or non-diseased) presenting to an Intermountain Healthcare facility.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2067-10-24 (Estimated); Study Completion 2077-10-24 (Estimated)

PRIMARY OUTCOMES:
Biobank for precision genomics | Day 0
  There are no primary endpoints planned for this biobank and endpoints will be specific to future research hypotheses. Investigators anticipate examining genetic and genomic data using a variety of molecular and cellular analysis techniques and in various tissues and fluids.
Biobank for precision transcriptomics | Day 0
  There are no primary endpoints planned for this biobank and endpoints will be specific to future research hypotheses. Investigators anticipate examining transcriptomic data using a variety of molecular and cellular analysis techniques and in various tissues and fluids.
Biobank for precision proteomics | Day 0
  There are no primary endpoints planned for this biobank and endpoints will be specific to future research hypotheses. Investigators anticipate examining proteomic data using a variety of molecular and cellular analysis techniques and in various tissues and fluids.

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Healthcare, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No